CLINICAL TRIAL: NCT03707730
Title: A Randomized, Double-Blind, Placebo Controlled, Crossover Trial to Evaluate Safety and Efficacy of AGY in Persons With Celiac Disease Age > 10 Years
Brief Title: A Randomized, Double-Blind, Placebo Controlled, Crossover Trial to Evaluate Safety and Efficacy of AGY in Celiac Disease
Acronym: AGY-010
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Igy Inc. (Industry)
Collaborators: Vetanda Group Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AGY-010
Record Dates: First submitted 2018-10-12; First posted 2018-10-16 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Celiac Disease
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Intervention Model Description: randomized double-blind, placebo-controlled crossover trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: placebo controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AGY (Experimental): capsule containing egg yolk with AGY
  Interventions: Dietary Supplement: AGY
- placebo (Placebo Comparator): capsule containing plain egg yolk
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: AGY — oral AGY taken prior to meals
  Arms: AGY
Other: placebo — oral placebo taken prior to meals
  Arms: placebo

SUMMARY:
To assess the efficacy and safety of AGY vs placebo when administered to individuals age 10 to 65 years with medically proven CD and on a gluten free diet

DETAILED DESCRIPTION:
We propose to conduct a randomized double-blind, placebo-controlled crossover trial in 149 individuals with celiac disease proven by biopsy (or other medically documented confirmation of CD, e.g. TTG counts > 10 times the upper limit of normal on two occasions) at least 12 months before study entry, and who are following a gluten-free diet but continue to have recurrent symptoms.

AGY is designed to neutralize the hidden gliadin in food, thus preventing gliadin absorption and gliadin induced pathogenesis. The study will test whether AGY is safe and effective in the study population, versus placebo.

Primary Objective: The primary objective will be to evaluate the effect of AGY on celiac symptoms using the daily Celiac Symptom Index (CSI).

Secondary objectives: Secondary objectives will be to evaluate product safety and the effect of AGY on quality of life, autoantibodies, and gut permeability.

ELIGIBILITY:
Inclusion Criteria:

* history of CD
* experience periodic celiac related symptoms
* following a gluten free diet for at least 12 months

Exclusion Criteria:

* severe complications of CD or chronic active GI disease
* type 1 diabetic
* pregnant or breast feeding
* daily ASA/NSAID use
* any condition that in the opinion of the investigator, would preclude safe participation

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2019-10-29 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
symptoms | 14 weeks
  celiac related symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Justine Turner, MD, PhD, Principal Investigator — University of Alberta
Locations (2):
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - St Boniface Hospital, Winnipeg, Manitoba

IPD SHARING:
Plan to Share IPD: No